CLINICAL TRIAL: NCT03216421
Title: Locoregional Breast Cancer Recurrence Following Targeted Intraoperative Radiotherapy (IORT) for Ductal Carcinoma in Situ (DCIS)
Brief Title: Intraoperative Radiation Therapy (IORT) in DCIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eileen Connolly, Assistant Professor, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAQ7853
Record Dates: First submitted 2017-07-11; First posted 2017-07-13 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
Keywords: DCIS; Intraoperative Radiation (IORT); Lumpectomy; Breast Conserving Surgery
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low/Intermediate Grade DCIS (Other): Subjects with Low/Intermediate Grade DCIS will complete quality of life questionnaires before and after the IORT.
  Interventions: Other: Quality of Life Questionnaires
- High Grade DCIS (Other): Subjects with High Grade DCIS will complete quality of life questionnaires before and after the IORT.
  Interventions: Other: Quality of Life Questionnaires

INTERVENTIONS:
Other: Quality of Life Questionnaires — Quality of Life questionnaires will be completed by each subject.

SUMMARY:
The goal of this study is to examine the role of Intraoperative Radiotherapy (IORT) in Ductal Carcinoma In-Situ (DCIS) and to improve the understanding of the clinical, radiographic, and patient-related impact of adopting IORT.

DETAILED DESCRIPTION:
With advances in technology and screening, the overdiagnosis and overtreatment of ductal carcinoma in situ (DCIS) have increased. Minimizing treatment toxicity and cost is a high priority area of research. Intraoperative Radiation Therapy (IORT)is a form of radiation where a single high dose of irradiation is applied to the tumor bed at the time of lumpectomy. Its use has not been previously studied in DCIS. Proposed advantages include decreased toxicity to adjacent tissue and organs, reduction in healthcare costs, and improved quality of life. The investigators hypothesize that IORT is a safe and patient-friendly alternative to whole breast irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed DCIS of the breast
* Clinical ≤ 3.0 cm unifocal lesion
* No clinical or pathological evidence of nodal involvement
* Operable DCIS, suitable for breast conserving surgery
* Plans to administer irradiation to the breast only
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3, however grade 4 patients may be enrolled at the discretion of the treating radiation oncologist
* Must have had a diagnostic mammogram or MRI performed within last 6 months
* Women of child-bearing potential must have a negative pregnancy test in accordance to institutional guidelines
* Women of child-bearing potential must agree to use adequate contraceptive precautions (defined as oral contraceptives, intrauterine devices, surgical contraceptives, or combination of condom and spermicide) from the time of negative pregnancy test through the radiation treatment period.
* English or Spanish speaking
* Able to sign informed consent
* Amenable to regular follow-up (according to research policies) for at least 5 years.

Exclusion Criteria:

* Histologic or clinical evidence of invasive breast cancer
* Multicentric cancer in the ipsilateral breast as diagnosed by clinical examination, imaging, or pathologic assessment, not amenable to excision with negative margins with a single lumpectomy
* Synchronous bilateral breast cancer at the time of diagnosis
* Pathologic or imaging evidence of lymph node involvement
* Any severe concomitant disease that may limit their life expectancy to less than 5 years.
* Prior history of breast cancer or in-field radiation in the ipsilateral breast.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of local recurrence | 5 years
  Defined by ipsilateral breast tumor recurrence

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Determine incidence of any distant or local recurrence after the breast-conserving surgery (BCS) and IORT
Overall survival | 5 years
  Quantify the overall survival in women with DCIS following BCS and IORT at 5 years.
Acute Toxicities associated with IORT | 6 months
  Quantify the frequency of acute toxicities that occur within 6 months of having BCS and IORT. Measured using physician and patient reported toxicity surveys.
Longterm radiation toxicity | 5 years
  Quantify the frequency of toxicities that occur at greater than 6 months after having BCS and IORT. Measured using using physician and patient reported toxicity surveys as well as photographic assessment of cosmetic outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Connolly, MD, Principal Investigator — Assistant Professor of Radiation Oncology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No